CLINICAL TRIAL: NCT04429464
Title: AcQBlate Force Confirmatory Study for Atrial Arrhythmias (AcQBlate Force-PRA)
Brief Title: AcQBlate Force Confirmatory Study for Atrial Arrhythmias
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restrictions related to COVID the sponsor has decided not to move forward with this study
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-14
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Atrial Arrhythmias
Keywords: ablation; atrial arrhythmia

STUDY DESIGN:
Intervention Model Description: The patient population will consist of men and women between the ages of 18 - 80 years, presenting for a de novo or repeat left-sided atrial ablation for symptomatic paroxysmal atrial fibrillation (PAF) or persistent atrial fibrillation (PerAF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Non-randomized (Experimental): All subjects will be treated using the Acutus Medical's AcQBlate Force Sensing Ablation Catheter in combination with the Qubic Force Sensing Module (AcQBlate Force Sensing System) to treat their arrhythmia.
  Interventions: Device: AcQBlate Force Sensing Ablation Catheter

INTERVENTIONS:
Device: AcQBlate Force Sensing Ablation Catheter — Confirmation that the AcQBlate Force System is safe and effective for the treatment of atrial arrhythmias

SUMMARY:
AcQBlate Force Confirmatory Study for Atrial Arrhythmias (AcQBlate Force-PRA)

DETAILED DESCRIPTION:
Acutus Medical's AcQBlate Force Ablation Catheter when used in combination with the Qubic Force Sensing Module (AcQBlate Force System), is indicated for cardiac electrophysiological mapping, delivery of diagnostic pacing stimuli, and radiofrequency ablation of sustained or recurrent atrial arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 to 80 years at time of consent.
* Clinically indicated and scheduled for a de novo or repeat catheter ablation of PAF or PerAF
* Willing and able to provide written informed consent to to participate in the study and agree to comply with all follow-up visits and evaluations for the duration of the study.

Exclusion Criteria:

* In the opinion of the investigator, any contraindication to the planned atrial ablation, including anticoagulation contraindications or sepsis
* Continuous AF > 12-months (long-standing persistent AF)
* Atrial arrhythmias secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiac cause.
* An implanted pacemaker or Implantable Cardiac Defibrillator (ICD).
* Structural heart disease or cardiac history as described below:
* Left ventricular ejection fraction (LVEF) < 35% based on transthoracic echocardiogram (TTE) within the previous 180-days.
* Left atrial size > 55 mm based on TTE within the previous 180-days.
* Evidence of heart failure (NYHA Class III or IV).
* Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for coronary artery bypass).
* Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve.
* Coronary artery bypass graft (CABG) or coronary angioplasty (PTCA) procedure within the last 90-days.
* Unstable angina or ongoing myocardial ischemia.
* Severe uncontrolled systemic hypertension (systolic pressure > 240 mm Hg, diastolic pressure > 140 mm Hg recorded within the last 30-days.
* Moderate or severe tricuspid stenosis or regurgitation.
* Moderate or severe mitral stenosis or regurgitation.
* Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder.
* Presence of a left atrial appendage occlusion device.
* Previous PV stenting or evidence of PV stenosis
* Body Mass Index (BMI) >40 kg/m2
* History of blood clotting or bleeding disease.
* Any prior history of documented cerebral infarct or systemic embolism (excluding post- operative deep vein thrombosis (DVT)).
* Pregnant or lactating (current or anticipated during study follow up).
* Current enrollment in any other study protocol where testing or results from the study may interfere with the procedure or outcome measurements for this study.
* Any other condition that, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Subjects that demonstrate electrical isolation of the intended ablation | At the end of their ablation procedure
  The Primary Endpoint for Performance is an analysis of the proportion of subjects that demonstrate electrical isolation (block) of the intended ablation targets.
Proportion of subjects who are free from device/procedure related Major Adverse Events | Through 30-days post procedure
  The Primary Endpoint for Safety is an analysis of the proportion of subjects who are free from device/procedure related Major Adverse Events (MAEs) that occur following the ablation procedure through 30-days.

SECONDARY OUTCOMES:
Subjects with freedom from an atrial arrhythmia | 30-days post index procedure
  The Secondary Endpoint for Performance is documentation of subjects with freedom from an atrial arrhythmia at 30-days post index procedure.
Analysis of all identified SAEs, SADEs, and UADEs. | Through 30-days post procedure
  The Secondary Endpoint for Safety is a recording and analysis of all identified serious adverse events (SAEs), serious adverse device effects (SADEs), and unanticipated adverse device effects (UADEs) through 30-days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia